CLINICAL TRIAL: NCT00852007
Title: A Phase I/II Study Evaluating the Safety and Efficacy of Vaccination With Autologous Dendritic Cells Loaded With Tn-MUC1 Peptide in Patients With Non-Metastatic Androgen Independent Prostatic Adenocarcinoma.
Brief Title: A Study Evaluating Vaccination of Prostate Cancer Patients With Self Dendritic Cells Expressing MUC1
Acronym: MUC1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CAN-ONC-001 CAN
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; dendritic cells; MUC-1; immune therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC-Tn-MUC (Experimental): DC-Tn-MUC1: autologous dendritic cells expressing Tn-MUC1. 1.2 x 10e7 dendritic cells per dose. 5 administrations (doses)may be given in total.
  Interventions: Biological: DC-Tn-MUC1: autologous dendritic cells expressing Tn-MUC1

INTERVENTIONS:
Biological: DC-Tn-MUC1: autologous dendritic cells expressing Tn-MUC1 — 1.2 x 10e7 dendritic cells per dose. One dose delivered intradermally (i.d.) and into a node (i.n.). Two weeks after this,two injections i.d. 2 weeks apart. Optional booster injections at 6 (i.d. and i.n.) and and 12 months (i.d.).

SUMMARY:
This study investigates the use of the patients own immune cells to treat prostate cancer. Cells are taken from the patient and grown in the laboratory to become specialized immune cells called dendritic cells. Dendritic cells instruct other immune cells to recognize and attack foreign substances such as bacteria, viruses, or abnormal proteins on cancer cells. A protein called Tn-MUC-1 is added to the cells.This protein is present on prostate cancer cells. The modified cells are injected back into the patient, with the intention that the dendritic cells will instruct other immune cells to attack the prostate cancer cells.

DETAILED DESCRIPTION:
Patients undergo one standard apheresis to harvest peripheral mononuclear cells for dendritic cell vaccine preparation. The modified cells (vaccine) are frozen so that multiple injections may be given. Patients my receive up to 5 injections. The vaccine is given either intradermally or into a lymph node.

Patients will undergo blood sample collection for immune response studies on the day of treatment and 2 weeks following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a histologically documented diagnosis of prostate cancer
* Subject was surgically castrated at least 3 months prior to study inclusion or has been pharmacologically castrated for a minimum of 3 months prior to study inclusion.
* Subject must meet one of the following PSA criteria:

  * A PSA value of ≥20ng/mL (µg/L) obtained 12 months prior to study inclusion OR
  * A 50% rise in PSA values with a minimum rise of 1.0 ng/ml (µg/L), within 6 months prior to study inclusion OR
  * A rise in PSA defined by 2 sequential increases in PSA values. inclusion. There must be at least 2 weeks between each qualifying PSA value.
* Subjects who have received anti-androgen therapy must have a documented withdrawal period prior to study inclusion.
* For a subject who has withdrawn from anti-androgen therapy LESS than 6 months prior to study inclusion, one of the following criteria is ALSO required for eligibility:

  * Following the completion of the anti-androgen withdrawal period, one post-withdrawal PSA value must be higher than the last pre-withdrawal PSA value OR
  * Following the completion of the anti-androgen withdrawal period, if the subject's PSA value decreased, then he can still qualify if two increases in PSA values (as described in 4c) are documented after post-withdrawal nadir.
* At the time of screening the subject has no distant metastatic disease.

Exclusion Criteria:

* Subject is less than 19 years of age.
* Subject has a PSA value < 1.0 ng/mL at screening
* Subject currently has evidence of distant metastases.
* Subject has not, in the opinion of the investigator, a life expectancy greater than 12 months.
* Subject has a local recurrence and is a candidate for local salvage therapy
* Subject having previously received therapy [including radiation, steroids, radionuclides (such as rhenium, strontium or samarium), cryotherapy or cytotoxic chemotherapy] for prostate cancer are ineligible as defined below:

  * Subjects who received previous cytotoxic chemotherapy or radionuclide therapies are ineligible
  * Subjects who received therapy to the prostatic bed (external beam radiotherapy, brachytherapy or cryotherapy) within 6 months prior to study entry are ineligible.
  * Subjects who received radiation therapy to any lesion outside the prostate bed more than 6 months after castration or hormone initiation are ineligible.
  * Subjects who received steroids for the treatment of prostate cancer within 6 months prior to study entry are ineligible.
* Subjects having previously received opioid analgesic therapy.
* Subjects has received any of the following within 4 weeks of study entry:

  * Cyproterone acetate, ketoconazole, PC-SPES or other hormonally active therapies (with the exception of GnRH agonists or antagonists).
  * An investigational product
* Subject is on a concurrent steroids or immunosuppressive therapy for chronic inflammatory disease.
* Subject has had other malignancies within the previous 5 years with the exception of non-melanoma skin cancer.
* Subject has a score >1 on the ECOG Performance Scale (see Appendix I)
* Subject has an inadequate hematologic function
* Subject has inadequate liver function.
* Subject has a creatinine clearance <40 mL/min
* Subject has a known history of cardiovascular disability status of New York Heart Association Class ≥2.
* Subject has a history of uncontrolled asthma
* Subject has autoimmune disease(s)
* Subject has active infection(s)
* Subject is receiving antiretroviral therapy.
* Subject has received blood transfusion within 8 weeks of study inclusion.
* Subject has a clinically significant, unstable, uncontrolled disease that could be adversely affected by study participation.
* Subject has known allergy to shellfish

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2014-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Time to radiographic progression | Time to radiographic progression defined as the time from the first treatment to the occurence of any metastatic disease
  Radiographic disease as measured by the occurence of any metastatic disease based on modified RECIST 1.0 and/or the appearance of 2 or more new lesions on a bone scan.

SECONDARY OUTCOMES:
Number of participants with adverse events | Ongoing up to 2 years
  Acute and late toxicities as assessed by NCI CTCAE v 4.0
Time to PSA progression | Up to 2 years
Immune response | Up to 2 years
  Immune response defined as the induction of a cellular (CD4/CD8)response measured by CFSE or ICS assay and/or the induction of a humoral response as measured by an increase in specific antibody or the occurence of antibody isotype switching.
Overall survival | Up to 2 years
Disease-specific survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre P. Major, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada